CLINICAL TRIAL: NCT00629330
Title: Dissemination of Prostate Cancer Screening to Primary Care Physicians in African American Communities
Brief Title: Dissemination of Prostate Cancer Screening to PCP's in African American Communities
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left the institution.
Sponsor: Columbia University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Theresa J. Miller, Ph.D., Grants Manager, United States Army Medical Research and Materiel Command (USAMRMC)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: AAAA6313; PC020492 (Other: Department of Defense)
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2011-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate cancer screening; prostate specific antigen; African American males
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-component Academic Detailing (Experimental): Includes an interactive, digitized CDROM, focused on the discussion of risks and benefits, screening options or alternatives, values clarification, and mutual decision-making, alongside patient education materials designed for low literacy patients.
  Interventions: Behavioral: Academic Detailing

INTERVENTIONS:
Behavioral: Academic Detailing — Multi-component academic detailing including an interactive, digitized CD-ROM, focused on the discussion of risks and benefits, screening options or alternatives, values clarification, and mutual decision-making, alongside patient education materials designed for low literacy patients
  Other Names: Multi-component Academic Detailing

SUMMARY:
The aims of this project are to adapt and extend the use of academic detailing to the dissemination of prostate cancer (CaP) screening findings to primary care physicians practicing in African American communities. The objectives of this study are:

1. To test the hypothesis that a community physician-based educational intervention (multi-component academic detailing, including an interactive, digitized, web-based program for informed decision-making about prostate cancer, and patient education materials designed for low literacy patients) will increase physician knowledge, positive attitudes/beliefs toward screening and screening options, and prostate cancer screening (using the digital rectal exam, and the serum prostate specific antigen test) at baseline, 6-, and 12-months post- randomization, compared to the rate observed in a service- as-usual control.

1A. To demonstrate the feasibility of disseminating the American Cancer Society guidelines for prostate cancer screening among primary care practitioners using multi-component academic detailing.

2. To develop models predicting which physician offices are most and least likely to adopt the intervention, and to generate hypotheses about tailoring the dissemination of PC screening guidelines to different physician subgroups.

The long term goal of this project is to increase prostate cancer screening among African American communities, thus decreasing cancer-related morbidity and mortality.

DETAILED DESCRIPTION:
We will conduct a two-arm trial, recruiting, obtaining consent, then assigning 200 physicians' offices at random to one of two arms: intervention (multi-component academic detailing including an interactive, digitized CD-ROM, focused on the discussion of risks and benefits, screening options or alternatives, values clarification, and mutual decision-making, alongside patient education materials designed for low literacy patients) or to a service-as-usual control arm. We will query 200 physicians about their PC knowledge, attitudes/beliefs toward screening and screening options, and PSA testing at baseline, 6, and 12months post-randomization, compared to the rate observed in a service-as-usual control. Physician counseling in cancer control will be verified by a chart review at baseline and at 12months post-randomization (N=750). The instruments will assess prostate cancer knowledge, attitudes and beliefs toward screening, and uptake of the PSA. The nested design uses the physician's office as the unit of randomization, and the office as the unit of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Charts of male patients age 45 -75, (using the average age of death in this population) with at least one visit to the primary care provider over the last two years will be reviewed.

Exclusion Criteria:

Exclusion criteria will include:

* Diagnosis of cancer other than non-melanotic skin cancer.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
PSA and DRE | 12-month followup

SECONDARY OUTCOMES:
Counseling on PSA testing | 12-month followup

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Sheinfeld Gorin, PhD, Principal Investigator — Columbia University